CLINICAL TRIAL: NCT02527486
Title: Airway Registry for Chronic Airway Diseases
Brief Title: Seoul National University Airway Registry
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chang-Hoon Lee, Associate professor, Seoul National University Hospital
Other Study IDs: AW_registry
Record Dates: First submitted 2014-12-19; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Asthma; Asthma With Chronic Obstructive Pulmonary Disease; Bronchiectasis; Inactive Tuberculosis of Lung; Chronic Obstructive Airway Disease
Keywords: COPD; Asthma; ACOS; Bronchiectasis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood (whole blood, serum, plasma, buffy coat) Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- No predefined subgroups

SUMMARY:
This is a multicenter, prospective observational cohort study, in which patients with chronic airway diseases including chronic obstructive pulmonary disease(COPD), asthma, asthma-COPD overlap syndrome (ACOS) will be recruited.

ELIGIBILITY:
COPD

Inclusion Criteria:

* Postbronchodilator FEV1/FVC < 0.7 AND chronic respiratory symptom

Exclusion Criteria:

-

Asthma

Inclusion Criteria:

* Never smoker or <5PY of smoking history AND Recurrent episodes of asthma symptoms (wheezing, dyspnea, chest tightness, cough) AND (either Positive BDR OR positive metacholine/mannitol/exercise provocation test)

Exclusion Criteria:

-

ACOS

Inclusion Criteria:

* COPD AND Asthma (regardless of smoking status)

Exclusion Criteria:

-

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD Asthma ACOS Bronchiectasis TB-destroyed lung Other chronic airway diseases
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2011-09; Primary Completion 2021-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Death (time to death) | upto 20 years
  death from any cause, death from COPD-specific cause, death from CVD, malignancy

SECONDARY OUTCOMES:
post-bronchodilator FEV1 change rates | upto 20 years (at least 3 years)

OTHER OUTCOMES:
Time to 1st exacerbation (definition of exacerbation is described below) | upto 20 years
  Definition of exacerbation: Airway disease symptom aggravation requiring either (1) Use of antibiotics or steroid, or (2) visiting ER or hospitalization
Annual rate of exacerbation (definition of exacerbation is described below) | upto 20 years
  Definition of exacerbation: Airway disease symptom aggravation requiring either (1) Use of antibiotics or steroid, or (2) visiting ER or hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Chul-Gyu Yoo, M.D., Study Chair — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Seoul Metropolitan Government-Seoul National University Boramae Medical Center, Seoul

REFERENCES:
- [Derived] Jo YS, Park S, Kim DK, Yoo CG, Lee CH. The cutoff point of clinical chronic obstructive pulmonary disease questionnaire for more symptomatic patients. BMC Pulm Med. 2018 Feb 27;18(1):38. doi: 10.1186/s12890-018-0601-0. PMID 29482616
- [Derived] Jo YS, Lee J, Yoon HI, Kim DK, Yoo CG, Lee CH. Different prevalence and clinical characteristics of asthma-chronic obstructive pulmonary disease overlap syndrome according to accepted criteria. Ann Allergy Asthma Immunol. 2017 Jun;118(6):696-703.e1. doi: 10.1016/j.anai.2017.04.010. PMID 28583262